CLINICAL TRIAL: NCT03418831
Title: Selective Estrogen Receptor Modulators - Adjunctive Treatment for Negative and Cognitive Symptoms of Schizophrenia in Postmenopausal Women
Brief Title: Adjunctive Selective Estrogen Receptor Modulators on Negative and Cognitive Symptoms of Schizophrenia in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-YJ-01
Record Dates: First submitted 2018-01-22; First posted 2018-02-01 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-02

CONDITIONS: Schizophrenia
Keywords: negtive symptoms; cognitive function
MeSH Terms: conditions — Schizophrenia | interventions — Raloxifene Hydrochloride; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Raloxifene (Active Comparator): Raloxifene Hydrochloride
  Interventions: Drug: Raloxifene Hydrochloride
- Placebo (Placebo Comparator): placebo tablet
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Raloxifene Hydrochloride — 60 mg per capsule (1 tablet daily) for 12 weeks
  Other Names: Evista
  Arms: Raloxifene
Other: Placebo — 1 tablet daily for 12 weeks
  Other Names: Starch capsule
  Arms: Placebo

SUMMARY:
The aim of the project is to assess the efficacy of Adjunctive Selective Estrogen Receptor Modulators (Raloxifene) on Negative and Cognitive symptoms of Schizophrenia in Postmenopausal Women.

For postmenopausal women with schizophrenia, current research suggests that these people can be treated with estrogen, which can reduce cardiovascular and reproductive tissue problems, help sleep and improve mood. In addition, cognitive problems in this group of people can also be helped. Raloxifene is a Selective Estrogen Receptor Modulator (SERM), which means that it can affect the central nervous system (CNS) effects of estrogen (eg. improving emotional symptoms, memory, information processing and concentration), without adversely affecting reproductive tissue/organs such as breast, uterus and ovaries. The investigators are conducting a double-blind, placebo controlled, 12 weeks study comparing the negative symptoms and cognitive functions in postmenopausal women with schizophrenia in both groups. One group will receive clozapine plus 60mg Raloxifene (Usage: take 60mg Raloxifene tablets half an hour after breakfast every day, that is, take 1 tablet a day), while the second group will receive clozapine plus oral placebo (Usage: take 1 placebo half an hour after breakfast every day).

Hypothesis 1: Adjuvant raloxifene therapy in postmenopausal women with schizophrenia can improve negative symptoms, as measured on the rating scales, compared with the women receiving adjunctive placebo.

Hypothesis 2: The cognitive function of postmenopausal female schizophrenic patients treated with raloxifene would be better than that of the placebo group.

Hypothesis 3: That the Raloxifene group has less adverse reactions in postmenopausal women with schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a mental illness with unknown cause and difficult treatment which the global lifetime prevalence rate of about 1%. The core symptoms of schizophrenia include positive symptoms, negative symptoms, and impairment of cognitive function. Positive symptoms in most patients after antipsychotic treatment can significantly alleviate after antipsychotic treatment, but negative symptoms and cognitive deficits persist. Unfortunately, the long-term prognosis and social function of patients mainly depend on the degree of the rehabilitation of negative symptoms and cognitive function. At present, clinical research domestic and overseas on the negative symptoms and cognitive function gradually increased, but end up with the poor consistency of research results. The reason is various, but in any case, improving the treatment strategy is still very important.

Epidemiological data suggest that the age of onset of female schizophrenia is later than men, most of which are onset abruptly, and females have higher susceptibility to mental illness and relapse during the two important periods with hormonal changes. The first is in the postpartum, menopause is the second. It may be related to the lack of estrogen function. Therefore, we believe that the onset and symptoms of some female patients with schizophrenia are related to the dysfunction of estrogen. Many studies abroad have found that estrogen and selective estrogen receptor modulators have significant effects on female patients with schizophrenia, especially on negative symptoms and cognitive functions, but the clinical application is limited due to the potential side effects of estrogen.

Raloxifene is the second generation of selective estrogen receptor modulator, for the prevention and treatment of osteoporosis in postmenopausal women, which can significantly reduce the incidence of vertebral fractures. The common adverse drug reaction is slight increase in hot flash and leg cramps, and the most serious adverse drug reaction is venous thromboembolism. Past research has found that raloxifene can reduce the risk of decline in memory and attention, and taking raloxifene helps sleep. Current research suggests that as an adjuvant therapy, it can improve symptoms of menopausal women with schizophrenia (emotional symptoms, memory, information processing and storage), and will not negatively affect reproductive tissues or organs, such as breast, uterus and ovary.

According to the domestic and overseas research results, and based on the theoretical background of schizophrenia in estrogen insufficiency, we proposed randomized double-blind placebo-controlled study, in order to understand the effect of raloxifene on negative symptoms and cognitive function in adjuvant treatment of menopausal female patients with schizophrenia, meanwhile assess the adverse reactions after the treatment, provide the basis for clinical treatment of schizophrenia patients with negative symptoms and cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient or inpatient, aged more than 45 years, postmenopausal female (menopause for more than one year)
2. International Classification of Diseases, Tenth Revision, diagnosis of schizophrenia
3. Continue to receive antipsychotic clozapine for more than 2 years with a stable dose of at least one month
4. Negative symptoms scale >20 in PANSS, and a score of 4 (moderate) or more on one or more of N1-N7, and within two weeks before intervention, the total score of negative symptom factors improved by no more than 10%
5. Able to give informed consent

Exclusion Criteria:

1. Participating in other clinical studies
2. Previous use of raloxifene intolerable
3. Hormone related endocrine disease
4. Acute liver disease
5. thrombotic disease
6. Estrogen dependent tumor
7. Hyperthyreosis
8. Severe cardiac dysfunction or renal disease
9. Diabetes mellitus
10. Abnormal uterine bleeding or cerebrovascular accident
11. Hormone replacement therapy
12. using mood stabilizer

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Response in negative symptoms | baseline, week 4, 8, 12
  A response in negative symptoms was defined as improvement of ≥20% compared with baseline PANSS negative score (12 weeks)

SECONDARY OUTCOMES:
Clinical Assessment Interview for Negative Symptoms(CAINS) | baseline, week 4, 8, 12
  The CAINS is a scale of the clinical assessment interview for negative symptoms of schizophrenia.The CAINS includes 16 items covering motivation and pleasure across social (five items), vocational (three items), and recreational life (three items) domains, as well as emotion expression and speech (five items).All items were rated on a scale of 0-4, with higher scores reflecting greater impairment.
Scale for the Assessment of Negative Symptoms (SANS) | baseline, week 4, 8, 12
  The SANS are the most widely used symptom rating scales in schizophrenia research. SANS Total (Composite) score = sum(of SANS items 1-7, 9-12, 14-16, 18-21, and 23-24).The total range is from 0-120 scores.
Repeatable Battery for the Assessment of Neuropsychological Status(RBANS) | baseline, week 12
  The RBANS is a brief cognitive screening battery consisting of 12 subtests which are used to create Index scores in the following five cognitive domains: Immediate Memory, Visuospatial/Constructional Skills, Language, Attention, and Delayed Memory. A total score is created by summing the five index cores which are thought to represent one's current neuropsychological status.
Hormone level change | baseline, week 4, 8, 12
  Hormone level change over study duration (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: LV QINYU, Principal Investigator — SHANGHAI MENTAL HEALTH CENTRE
Locations (1):
- CHINA, Shanghai, Minhang, China

IPD SHARING:
Plan to Share IPD: Undecided